CLINICAL TRIAL: NCT07084688
Title: Swiss Cardiovascular-Kidney-Liver-Metabolic (CKLM) Registry
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-00756; am25Vischer
Record Dates: First submitted 2025-07-08; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Cradiovascular-kidney-liver-metabolic (CKLM) Syndrome; Cardiovascular-kidney-metabolic Syndrome
Keywords: Cardiovascular-kidney-liver-metabolic (CKLM) syndrome; Cardiovascular disease (CVD); Chronic kidney disease (CKD); Organ-specific diseases; Cardiovascular-kidney-metabolic (CKM) syndrome
MeSH Terms: conditions — Syndrome; Cardiovascular Diseases; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this clinical and exploratory Swiss Cardiovascular-Kidney-Liver-Metabolic (CKLM) Registry is to establish high quality prevalence and incidence database for Cardiovascular-Kidney-Metabolic (CKM) syndrome, its major contributors, and the extent of the respective organ damaged.

DETAILED DESCRIPTION:
The Swiss Cardiovascular-Kidney-Liver-Metabolic (CKLM) Registry is a prospective, longitudinal, non-interventional registry based at the Medical Outpatient Department of the University Hospital Basel. It aims to address key knowledge gaps related to (I) the prevalence, incidence, and heterogeneity of CKLM syndrome and its clinical phenotypes, (II) liver involvement, (III) emerging therapies, and (IV) the need for interdisciplinary care and integrated management. The registry supports improved understanding and management of this complex syndrome in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Individuals diagnosed with cardiovascular-kidney-metabolic (CKM) syndrome stages 0 to 3 according to the American Heart Association (AHA) or liver disease defined by any of the following:

  * For stage 0: Individuals without overweight/obesity, metabolic risk factors (normoglycemia, normotension, normal lipid profile), Chronic kidney disease (CKD), or Cardiovascular disease (CVD)
  * Individuals with overweight/obesity or dysfunctional adipose tissue, without other metabolic risk factors or CKD
  * Individuals with metabolic risk factors (hypertriglyceridemia, arterial hypertension, metabolic syndrome, diabetes) or CKD
  * Subclinical Atherosclerotic cardiovascular disease (ASCVD) or subclinical heart failure (HF) in individuals with excess/dysfunctional adiposity, other metabolic risk factors, or CKD in the clinical assessment[2]
  * Independent of CKM syndrome stages, individual with signs of hepatic steatosis on imaging
* Willingness to provide informed consent

Exclusion Criteria:

* Individuals with CKM syndrome stage 4 according to the AHA

  * Individuals with clinical cardiovascular disease including:
  * History of coronary artery disease, myocardial infarction, coronary artery intervention
  * History of atrial fibrillation
  * History of stroke
  * Symptomatic peripheral artery disease (>stage I)
  * History of symptomatic HF
  * History of HF hospitalisation
* Inability to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 200-300 participants with cardiovascular-kidney-metabolic (CKM) syndrome per year at the Medical Outpatient Department of the University Hospital Basel
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-07-14 (Estimated); Primary Completion 2040-07 (Estimated); Study Completion 2040-07 (Estimated)

PRIMARY OUTCOMES:
Frequency of cardiovascular diseases | At baseline, 6, 12 months and annually up to 10 years
  Out of available clinical data from the local electronic health record the frequency of cardiovascular diseases (e.g. stroke, myocardial infarction, coronary artery disease, peripheral arterial disease, hypertension, heart failure) will be assessed
Frequency of kidney diseases | At baseline, 6, 12 months and annually up to 10 years
  Out of available clinical data from the local electronic health record the frequency of kidney diseases (e.g. chronic kidney disease, kidney failure) will be assessed
Frequency of liver diseases | At baseline, 6, 12 months and annually up to 10 years
  Out of available clinical data from the local electronic health record the frequency of liver diseases (e.g. Metabolic Dysfunction-associated steatotic liver disease, MASLD) will be assessed
Frequency of metabolic diseases | At baseline, 6, 12 months and annually up to 10 years
  Out of available clinical data from the local electronic health record the frequency of metabolic diseases (e.g. dyslipidemia, pre-/diabetes) will be assessed
Frequency of microalbuminuria | At baseline, 6, 12 months and annually up to 5 years
  Frequency of microalbuminuria
Frequency of increased HbA1c | At baseline, 6, 12 months and annually up to 5 years
  Frequency of increased HbA1c
Assessment of Fib4-score | At baseline, 6, 12 months and annually up to 5 years
  Assessment of Fib-4 score
Signs of hypertensive heart disease | At baseline, 6, 12 months and annually up to 10 years
  Signs of hypertensive heart disease at transthoracic echocardiography determined by left ventricular hypertrophy (LVH)
Signs of steatosis hepatis | At baseline, 6, 12 months and annually up to 5 years
  Signs of steatosis hepatis in abdominal sonography defined as increased liver echogenicity
Structured, registry specific questionnaire | At baseline and annually up to 10 years
  The structured questionnaire is register-specifically designed and focuses on questions related to health behavior, medical history, mental health disorders, social determinants of health and adverse events. The collected data are aggregated to allow for standardized evaluation of key domains across the study population.
EQ-5D-5L | At baseline and annually up to 10 years
  Assessment of quality of life with the EQ-5D-5L ( (European Quality of Life 5 Dimensions 5 Level Version) tool within the study specific questionaire. 5 Dimensions of quality of life will be asked and coded in a 1-digit number that describes health state. Higher 1-digit numbers indicate a worse outcome. The tool also includes a EQ visual analogue scale (VAS), a quantitative and subjective measure of health outcome. Higher values indicate a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Annina Vischer, PD Dr. med., Principal Investigator — Medical Outpatient Department and Hypertension Clinic, ESH Hypertension Centre of Excellence, University Hospital Basel
Locations (1):
- Medical Outpatient Department of the University Hospital Basel, Basel, Canton of Basel-City, Switzerland